CLINICAL TRIAL: NCT03209739
Title: Can a WhatsApp Reminder Improve the Quality of Screening Colonoscopy? A Randomized Controlled Study
Brief Title: WhatsApp Reminder on Bowel Preparation Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Nursing Officer, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: WhatsApp BPrep Study
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Bowel Preparation; WhatsApp Messenger; Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Endoscopists will be masked if the patients have received WhatsApp reminder prior colonoscopy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp reminder (Active Comparator): An additional WhatsApp reminder with same content of the written instruction and a video of explanation of bowel preparation by a nurse 4 days prior colonoscopy
  Interventions: Other: WhatsApp reminder
- No reminder (No Intervention): No additional reminder will be given

INTERVENTIONS:
Other: WhatsApp reminder — An additional WhatsApp reminder with same content of the written instruction and a video of explanation of bowel preparation by a nurse 4 days prior colonoscopy
  Arms: WhatsApp reminder

SUMMARY:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 2014.

CRC is one of the most preventable cancers because its development in general follows an adenoma-carcinoma sequence. Adenomas are considered precursor lesions for CRC. Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 50. Modalities such as guaiac-based fecal occult blood tests (gFOBT), fecal immunochemical tests (FIT), flexible sigmoidoscopy (FS), and colonoscopy are among the acceptable options for CRC screening.

While early detection and removal of colorectal adenoma by screening colonoscopy with polypectomy reduce CRC incidence and mortality, interval cancers (cancers that develop after a colonoscopy and before the next scheduled colonoscopy) may still occur and were reported to account for up to 10.5% of CRC. a CRC has been associated with proximal colon location, small lesion, flat lesion, missed lesion, inadequate examination, incomplete resection of lesion, tumor biology, and low adenoma detection rate (ADR). High ADR (eg, ≥ 20%) has been associated with a reduced risk of interval CRC.

Bowel preparation includes diet restriction and proper use of laxative before the colonoscopy, and this is one of the important factors to ensure a high quality colonoscopy. Suboptimal bowel preparation may lead to decreased ADR, cecal intubation rate, and surveillance interval and increased procedural time. Efforts to improve bowel cleansing quality through traditional communication routines, including face-to-face verbal education, written booklet or visual aids or telephone-based re-instruction have proven to be useful. A recent study using WeChat, a widely used social media mobile app in China, has also shown to be effectively improving bowel preparation level of a mixed population who received diagnostic (77%), screening (15.8%) and surveillance (7.2%) colonoscopy. However, the impact of social media mobile app on the bowel preparation level of screening colonoscopy is not yet known. Hence, this study will investigate the effectiveness of the most popular social media app worldwide, WhatsApp in bowel preparation level of screening colonoscopy.

DETAILED DESCRIPTION:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 2014.

CRC is one of the most preventable cancers because its development in general follows an adenoma-carcinoma sequence. Adenomas are considered precursor lesions for CRC. Recent guidelines from USA, Europe and Asia Pacific region recommend CRC screening for average-risk asymptomatic individuals starting at age 50. Modalities such as guaiac-based fecal occult blood tests (gFOBT), fecal immunochemical tests (FIT), flexible sigmoidoscopy (FS), and colonoscopy are among the acceptable options for CRC screening.

While early detection and removal of colorectal adenoma by screening colonoscopy with polypectomy reduce CRC incidence and mortality, interval cancers (cancers that develop after a colonoscopy and before the next scheduled colonoscopy) may still occur and were reported to account for up to 10.5% of CRC. a CRC has been associated with proximal colon location, small lesion, flat lesion, missed lesion, inadequate examination, incomplete resection of lesion, tumor biology, and low adenoma detection rate (ADR). High ADR (eg, ≥ 20%) has been associated with a reduced risk of interval CRC.

Bowel preparation includes diet restriction and proper use of laxative before the colonoscopy, and this is one of the important factors to ensure a high quality colonoscopy. Suboptimal bowel preparation may lead to decreased ADR, cecal intubation rate, and surveillance interval and increased procedural time. Efforts to improve bowel cleansing quality through traditional communication routines, including face-to-face verbal education, written booklet or visual aids or telephone-based re-instruction have proven to be useful. A recent study using WeChat, a widely used social media mobile app in China, has also shown to be effectively improving bowel preparation level of a mixed population who received diagnostic (77%), screening (15.8%) and surveillance (7.2%) colonoscopy. However, the impact of social media mobile app on the bowel preparation level of screening colonoscopy is not yet known. Hence, this study will investigate the effectiveness of the most popular social media app worldwide, WhatsApp in bowel preparation level of screening colonoscopy.

Subjects already recruited by other studies in Institute of Digestive Disease and arranged for an out-patient screening colonoscopy will be identified and recruited.

Demographic data including age, sex, smoking and alcohol habits, comorbidities, education level, family income, time of using WhatsApp of the eligible subjects will be collected. Subjects will then be randomized to either standard group or WhatsApp group. As a usual practice, all subjects will receive a verbal explanation of bowel preparation by a healthcare professional on the day of appointment making. A detailed written bowel preparation instruction will be also given to subjects.

For subjects randomized to the WhatsApp reminder group, they will receive an additional WhatsApp reminder with same content of the written instruction and a video of explanation of bowel preparation by a nurse 4 days prior colonoscopy. Subjects are encouraged to ask any question regarding the bowel preparation via WhatsApp. All these enquiries will be replied by the principal investigator during office hours.

The colonoscopy results, including, the bowel preparation level and the number and nature of lesion found (if any) will be collected afterwards. Two investigators reviewed all the colonoscopy videos independently to grade the quality of bowel preparation by Boston Bowel Preparation Scale.

ELIGIBILITY:
Inclusion Criteria:

* Subjects arranged for an out-patient screening colonoscopy in Prince of Wales Hospital and Alice Ho Miu Ling Hospital.

Exclusion Criteria:

* Lack of access to WhatsApp Messenger

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Bowel preparation level | Immediate after colonoscopy
  Proportion of subjects having optimal bowel preparation level

SECONDARY OUTCOMES:
Polyp detection rate | Immediate after colonoscopy
  Proportion of subjects having a polyp detected
adenoma detection rate | a month after colonoscopy
  Proportion of subjects having a adenoma detected
Mean number of adenoma detected per patient | 1 year after study started, i.e. when all subjects undergo colonoscopy
  Mean number of adenoma detected per patient

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yuen Tung Lam, MSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lam TYT, Wu PI, Tang RSY, Tse YK, Lau JYW, Wu JCY, Sung JJY. Nurse-led reinforced education by mobile messenger improves the quality of bowel preparation of colonoscopy in a population-based colorectal cancer screening program: A randomized controlled trial. Int J Nurs Stud. 2022 Sep;133:104301. doi: 10.1016/j.ijnurstu.2022.104301. Epub 2022 May 30. PMID 35764027